CLINICAL TRIAL: NCT04542473
Title: Pancreatic Enzymes and Bile Acids: A Non-Antibiotic Approach to Treat Intestinal Dysbiosis in Acutely Ill Severely Malnourished Children
Brief Title: Pancreatic Enzymes and Bile Acids in Acutely Ill Severely Malnourished Children
Acronym: PB-SAM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: University of Amsterdam (Other); University of Toronto (Other); University of Washington (Other); Oregon Health and Science University (Other); Kenya Medical Research Institute (Other); Queen Elizabeth Central Hospital, Blantyre, Malawi (Unknown); Makerere University (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OxTREC 43-20
Record Dates: First submitted 2020-08-06; First posted 2020-09-09 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: SEPSIS; MALNUTRITION, CHILD
Keywords: "small intestinal bacterial overgrowth"; "severe malnutrition"; "factorial"; "pancreatic enzymes"; "bile acids"; "bacterial"; "translocation"; "dysbiosis"; "inflammation"
MeSH Terms: conditions — Sepsis; Child Nutrition Disorders; Malnutrition; Dysbiosis; Inflammation | interventions — Pancrelipase; Ursodeoxycholic Acid

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized clinical trial 2x2 factorial design in 3 stages:
  In stage 1, (200 participants). Then the Data & Safety Monitoring Committee (DSMC) will review data for likelihood major safety signals/harm (non-inferior to placebo) based on a composite endpoint of toxicity, serious adverse events (SAEs) and deaths.
  In stage 2, (200 more participants, total 400 participants). Then the DSMC will review data on a composite endpoint of SAEs and deaths and results of modeled simulations for the likelihood of superiority over placebo for mortality. Interventions with less than 80% probability of efficacy will be discontinued. Sample size for stage 3 may be adjusted.
  In stage 3, (800 more participants, total target sample size 1,200) across all sites, based on a hazard ratio of 0.66 (a 33% reduction in mortality) from a baseline mortality of 24% to 16% with 90% power, 20% inflation for the factorial design and 5% loss to follow up.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sequential study numbers will be computer generated according to a blocked randomization list of random block sizes allocated to each site before the study begins.
  Identical study investigation medical product (IMP) packs will be labelled with sequential study numbers according to a prepared blocked randomization list before the trial begins. An independent off-site trial-pharmacist will implement labeling of the IMP with unique study numbers according to the randomization list.
  Study numbers will be issued in consecutive order at each site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pancreatic Enzymes (PE) (Active Comparator): Pancreatic enzymes formulated as 5000 IE lipase, 3600 IE amylase and 200 IE protease per 100 mg of granules, packaged as sachets. The target dose is 3000 IU lipase/kg, twice daily (1440 IU/kg amylase/80 IU/kg protease), which is the dose used for children with cystic fibrosis and exocrine pancreas insufficiency. For oedematous malnutrition, weight for dosing is reduced by 10%. To be prescribed following enrolment and given just prior to or during a feed. Prescription will follow weight bands to allow a lower range of 2000 IU/kg/day and upper range of 4000 IU/kg/day:
  Weight from Weight to Dose Dose Upper range Lower range (Kg) (Kg) (sachets) (IU Lipase) (IU/kg/dose) (IU Lipase)
  ---------------------------------------------------------------------------------------------------------- 2.50 4.99 2 10000 4000 2000 5.00 7.49 4 20000 4000 2670 7.50 9.99 6 30000 4000 3000 10.0 15.0 8 40000 4000 2667
  Interventions: Drug: Pancreatic Enzyme
- Placebo-PE (Placebo Comparator): Oral/enteral placebo matching active Pancreatic Enzymes (PE). Dose presentation in whole sachets of 100mg of granules. For oedematous malnutrition, weight for dosing is reduced by a pragmatic 10%. To be prescribed following enrolment and given just prior to or during a feed. Prescription will follow weight bands:
  Weight from Weight to Dose Dose Upper range Lower range (Kg) (Kg) (sachets) (IU Lipase) (IU/kg/dose) (IU Lipase)
  ----------------------------------------------------------------------------------------------------------------------------------------- 2.50 4.99 2 Nil Nil Nil 5.00 7.49 4 Nil Nil Nil 7.50 9.99 6 Nil Nil Nil 10.0 15.0 8 Nil Nil Nil
  Interventions: Other: Pancreatic Enzyme placebo
- Ursodeoxycholic acid (UA) (Active Comparator): The dose of ursodeoxycholic acid will be given at 10 mg/kg twice per day just prior to or during a feed, using a suspension of 50 mg/ml = 0.2 ml/kg. For oedematous malnutrition participants, weight is pragmatically reduced by 10%. To be prescribed and given following enrolment.
  Interventions: Drug: Ursodeoxycholic acid
- Placebo-UA (Placebo Comparator): The dose of placebo will be given twice per day just prior to or during a feed at 0.2 ml/kg. To be prescribed and given following enrolment.
  Interventions: Other: Ursodeoxycholic acid placebo

INTERVENTIONS:
Drug: Pancreatic Enzyme — CREON micro 5000
  Other Names: CREON
  Arms: Pancreatic Enzymes (PE)
Drug: Ursodeoxycholic acid — Ursodiol C24H40O4 suspension
  Other Names: UDCAMENT
  Arms: Ursodeoxycholic acid (UA)
Other: Pancreatic Enzyme placebo — Microcrystalline Cellulose,Macrogel 4000, Iron Oxide Yellow, Iron Oxide Red, Activated Charcoal.
  Other Names: Placebo-PE
  Arms: Placebo-PE
Other: Ursodeoxycholic acid placebo — Sodium Citrate Dihydrate, Aspartame, Carboxymethylcellulose Sodium, Citric Acid Monohydrate, Dispersible Cellulose, Glycerol, Polysorbate-80, Saccharin Sodium,Sodium Benzoate, Sodium Methylparaben, Sodium Propylparaben
  Other Names: Placebo-UA
  Arms: Placebo-UA

SUMMARY:
Children with severe malnutrition who are sick and admitted to hospitals have high mortality, usually because of infection. Malnourished children have more potentially harmful bacteria in their upper intestines than well-nourished children and this may contribute to inflammation in the gut and whole body. These bacteria may cross from the intestines to the bloodstream causing life-threatening infections. A related abnormality among malnourished children is reduction in the digestive enzymes made by the pancreas and the liver. Apart from helping with digestion of food, these enzymes are important in helping the body control bacteria in the upper intestines. It is therefore possible that treatment with digestive enzymes could help reduce the burden of harmful bacteria and thus lower inflammation and the risk of serious infection. One study conducted in Malawi has shown that children with severe malnutrition who were supplemented with pancreatic enzymes had a lower risk of dying. However, this was a small study and although promising, requires validation. No studies of supplementation with bile acids have been done among severely malnourished children. However, bile acids are commonly used to manage patients with liver function abnormalities, something that malnourished children suffer from as well. The investigators want to find out if supplementing these pancreatic enzymes and bile acids among ill children with severe acute malnutrition is safe and reduces the risk of death, deterioration or readmission to hospital.

DETAILED DESCRIPTION:
Severely malnourished children who present with an acute illness have a high risk of mortality. Severe malnutrition is associated with intestinal inflammation and changes in the fecal microbiome ('dysbiosis'). Apart from in the large intestine, dysbiosis is also present in the small (upper) intestine, where increased bacterial density and altered microbial composition can contribute to intestinal inflammation and intestinal dysfunction which may ultimately contribute to the development of sepsis and death. The bacterial density and composition in the small intestine can be altered using antibiotics. However, apart from side effects, antibiotic use contributes to the development of antibiotic resistance, which is very common in hospitalized malnourished patients and can pose a threat to both individual and public health. In addition to intestinal dysbiosis and intestinal inflammation, children with severe malnutrition suffer from impaired exocrine pancreatic and hepatobiliary function, which are important for nutrient digestion and absorption to aid their recovery.

One previous pilot trial showed that treating children with severe malnutrition with pancreatic enzymes led to a reduction in mortality. The investigators hypothesize that supplementing these enzymes exogenously to severely malnourished children will improve their clinical outcome by reducing dysbiosis, intestinal inflammation and sepsis.

The objective of this study is to determine whether treating ill severely malnourished children with pancreatic enzymes or bile acids is safe and improves mortality. The investigators will conduct a double blind, randomized clinical trial in a 2x2 factorial design in hospitalized severely malnourished children. Participants will be treated with pediatric formulations of pancreatic enzymes, bile acids, both or placebo for 21 days. Participants will be followed up daily during their hospital stay and on day 21 and 60 after enrollment.

This trial will be conducted in three stages to allow for careful interim evaluations to assess safety and study progress. After the first and second stage, interim analyses assess safety and likelihood of benefit before enrolling the full sample size to assess mortality as the primary outcome. Secondary outcomes include adverse events, length of hospital stay and growth. Exploratory outcomes will examine intestinal and systemic inflammation and metabolic changes to examine mechanisms affected by the interventions, and costs.

Two sub-studies will be conducted. In Kenya and Bangladesh, daily blood gases, lactate and biochemistry for the first 5 days to assess early clinical progress. In Malawi and Uganda, hydrogen breath testing will be used to evaluate impact on upper small intestinal bacterial overgrowth.

Overall, this trial will determine whether a non-antibiotic, bactericidal intervention given in additional to standard of care management reduces mortality in acutely ill severely malnourished children.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to <59 months
* Admitted to hospital with an acute, non-traumatic illness and within 72 hours of admission at the time of enrolment
* Severe malnutrition (weight-for-height <-3 z scores of the median WHO growth standards and/or mid upper arm circumference <115mm (<110mm age below 6 months), or symmetrical oedema of at least the feet related to malnutrition (not related to a primary cardiac or renal disorder)
* Able to feed orally in usual state of health.
* Accompanied by care provider who provides written informed consent
* Primary caregiver plans to stay in the study area during the duration of the study
* Presence of two or more features of severity as specified below. If a child meets two criteria, they may be enrolled before further criteria are assessed (e.g. a child may be eligible on clinical signs before the complete blood count results are known):

Respiratory distress "Subcostal indrawing" or "nasal flaring" or "head-nodding" Oxygenation "Central cyanosis" or SaO2 <90% Circulation Limb temperature gradient or capillary refill >3 seconds Conscious level AVPU < "A" Pulse > 180 per min Haemoglobin < 7g/dl Blood glucose < 3mmol/L White blood cells < 4 or > 17.5 x 109/L Temperature <36 or >38.5oC Very low MUAC MUAC <11cm

Exclusion Criteria:

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 60 days
  Death

SECONDARY OUTCOMES:
Rate of SAEs | 60 days
  All serious adverse events
Rate of toxicity events | 21 days
  Grade 3 or 4 toxicity events whilst receiving investigational products
Intestinal function | 60 days
  number of days with diarrhoea during index hospital admission
Antimicrobials | 60 days
  Days on second and third-line antibiotics during index admission and readmission
Hospitalisation duration | 60 days
  Number of days from enrolment to discharge during index admission
Growth - arm circumference cm | 60 Days
  Change in MUAC in cm between enrolment and 60 days later
Growth - weight for age z score | 60 days
  Change in weight for age z score between enrolment and 60 days later
Growth - weight for length z score | 60 days
  Change in weight for length z score between enrolment and 60 days later
Growth - length for age z score | 60 days
  Change in length for age z score between enrolment and 60 days later

CONTACTS AND LOCATIONS:
Overall Officials: James A Berkley, MD, Study Chair — University of Oxford
Locations (4):
- ICDDR,B Dhaka Hospital, Dhaka, Bangladesh
- KEMRI WT Clinical Trials Facility, Kilifi, Kenya
- Queen Elizabeth Central Hospital, Blantyre, Malawi
- Mulago Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
Anonymised data may be shared through application to DGC@kemri-wellcome.org. Datasets will be uploaded on the HARVARD DATAVERSE for managed access

REFERENCES:
- [Background] Zhang L, Voskuijl W, Mouzaki M, Groen AK, Alexander J, Bourdon C, Wang A, Versloot CJ, Di Giovanni V, Wanders RJ, Bandsma R. Impaired Bile Acid Homeostasis in Children with Severe Acute Malnutrition. PLoS One. 2016 May 10;11(5):e0155143. doi: 10.1371/journal.pone.0155143. eCollection 2016. PMID 27163928
- [Background] Bartels RH, Bourdon C, Potani I, Mhango B, van den Brink DA, Mponda JS, Muller Kobold AC, Bandsma RH, Boele van Hensbroek M, Voskuijl WP. Pancreatic Enzyme Replacement Therapy in Children with Severe Acute Malnutrition: A Randomized Controlled Trial. J Pediatr. 2017 Nov;190:85-92.e2. doi: 10.1016/j.jpeds.2017.07.013. Epub 2017 Sep 11. PMID 28912050
- [Background] Njunge JM, Gwela A, Kibinge NK, Ngari M, Nyamako L, Nyatichi E, Thitiri J, Gonzales GB, Bandsma RHJ, Walson JL, Gitau EN, Berkley JA. Biomarkers of post-discharge mortality among children with complicated severe acute malnutrition. Sci Rep. 2019 Apr 12;9(1):5981. doi: 10.1038/s41598-019-42436-y. PMID 30979939
- [Background] Attia S, Versloot CJ, Voskuijl W, van Vliet SJ, Di Giovanni V, Zhang L, Richardson S, Bourdon C, Netea MG, Berkley JA, van Rheenen PF, Bandsma RH. Mortality in children with complicated severe acute malnutrition is related to intestinal and systemic inflammation: an observational cohort study. Am J Clin Nutr. 2016 Nov;104(5):1441-1449. doi: 10.3945/ajcn.116.130518. Epub 2016 Sep 21. PMID 27655441
- See also: The CHAIN Network — http://www.chainnetwork.org